CLINICAL TRIAL: NCT00596791
Title: Ocular Signs and Symptoms in Glaucoma Patients Switched From Latanoprost 0.005% to Preservative Free Tafluprost Eye Drops
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Santen Oy (Industry)
Responsible Party: Auli Ropo, Study Director, Santen Oy
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Santen-77552; EudraCT number 2007-004872-37
Record Dates: First submitted 2008-01-08; First posted 2008-01-17 (Estimated); Last update posted 2009-01-12 (Estimated); Status verified 2009-01

CONDITIONS: Ocular Hypertension; Open-Angle Glaucoma
MeSH Terms: conditions — Ocular Hypertension; Glaucoma, Open-Angle | interventions — tafluprost

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 arm (Other): Open-lable study with one arm.
  Interventions: Drug: tafluprost

INTERVENTIONS:
Drug: tafluprost — prostaglandine analoque

SUMMARY:
The purpose of this study is to investigate if changes in ocular signs and symptoms occur in patients with ocular hypertension or glaucoma when they switch from latanoprost 0.005% (Xalatan) to preservative free Tafluprost eye drops.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of ocular hypertension or open angle glaucoma for which the patient has been using latanoprost 0.005% as his/her prior medication. - Evaluable patients must have ocular surface related symptoms and/or signs with their prior medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2008-01; Primary Completion 2008-07 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Change from screening in ocular symptoms and signs | at week 6 and 12

SECONDARY OUTCOMES:
Safety and Quality of life parameters. | From Screening (visit 1) to visits at week 2, 6 and 12.

CONTACTS AND LOCATIONS:
Overall Officials: Hannu Uusitalo, Professor, Principal Investigator — Finn-Medi Research, Finland
Locations (1):
- Finn-Medi Research Oy, Tampere, Finland